CLINICAL TRIAL: NCT04626908
Title: Clinical Study of Targeting CD19 and CD22 Chimeric Antigen Receptor T Lymphocytes in the Treatment of Recurrent or Refractory B Cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Huang (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC022F-ZhejiangU
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Relapsed and Refractory; Lymphoid Hematological Malignancies
Keywords: lymphoid hematological malignancies; CAR-T cell therapy; CD19; CD22
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of GC022F CAR-T cells (Experimental): Each subject receive GC022F CAR T-cells by intravenous infusion
  Interventions: Drug: GC022F CAR-T cells

INTERVENTIONS:
Drug: GC022F CAR-T cells — Each subject receive GC022F CAR-T cells by intravenous infusion
  Other Names: GC022F CAR-T cells injection

SUMMARY:
Clinical Study of Targeting CD19 and CD22 Chimeric Antigen Receptor T Lymphocytes in the Treatment of Recurrent or Refractory B Cell Non-Hodgkin Lymphoma

DETAILED DESCRIPTION:
This is a single-arm, single-center, open clinical study to evaluate the safety and efficacy of GC022F injection in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years old (including the threshold value);
2. Histologically confirmed as diffuse large B-cell lymphoma (DLBCL), transformed follicular lymphoma (TFL), or primary mediastinal B-cell lymphoma (PMBCL) :

   i. Refractory B-NHL: PD was the optimal response to standard first-line treatment (those with intolerance to first-line treatment were not included in this study); Or SD after at least 4 courses of first-line treatment, and the DURATION of SD shall not exceed 6 months after the last treatment; Or the subjects' best response to the last treatment of second-line or above treatment is PD, or SD after at least 2 courses of second-line or above treatment, and the SD maintenance time is not more than 6 months; Or:

   ii. Relapsed B-NHL: after standard systemic treatment and complete remission after second-line treatment, the disease recurred as certified by histopathology, or the recurrence as confirmed by histopathology within 1 year after autologous hematopoietic stem cell transplantation (not limited by previous treatment methods);

   iii. Patients with INVERt follicular lymphoma must receive chemotherapy prior to transformation and meet the above definition of recurrent or refractory after transformation;
3. according to Lugano treatment response standard (2014 version), there should be at least one evaluable tumor lesion: the longest diameter of the injunctional lesion was > 1.5cm, and the longest diameter of the injunctional lesion was b> 1.0cm;
4. Positive expression of CD19 and CD22 in biopsy sections of tumor tissues;
5. Patients who have failed or relapsed after single-target CAR-T therapy may also be enrolled.
6. Prior to the study, the approved anti-B-NHL treatment, such as systemic chemotherapy, general radiotherapy and immunotherapy, has been completed for at least 2 weeks;
7. ECOG≤1；
8. Expected survival ≥3 months;
9. Absolute count of neutrophils ≥ 1×109/L;
10. Platelet count ≥50×109/L;
11. Absolute lymphocyte count ≥1×108/L;
12. Adequate organ function reserve:

    1. ALANINE aminotransferase and aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value);
    2. Creatinine clearance rate (Cockcroft-Gault method) ≥60 mL/min;
    3. Serum total bilirubin ≤1.5× UNL;
    4. The left ventricular ejection fraction (LVEF) of the subject was diagnosed by echocardiography ≥50%, and no clinically significant pericardial effusion was observed, and no clinically significant ecg abnormalities were observed;
    5. under natural indoor air environment, the basic oxygen saturation of > is 92%;
13. Vein access required for collection can be established, and there are no contraindications for leukocyte collection;
14. Women of childbearing age had negative pregnancy test during screening period and before administration, and agreed to take effective contraceptive measures at least one year after infusion; male subjects with fertile partners must agree to use effective barrier contraceptive method at least one year after infusion and avoid sperm donation;
15. Voluntary signing of informed consent.

Exclusion Criteria:

1. Other tumors (except cured non melanoma skin cancer, cervical cancer in situ, superficial bladder cancer, breast ductal carcinoma in situ, or other malignant tumors with complete remission for more than 5 years);
2. Persons with severe mental disorders;
3. A history of hereditary diseases such as Fanconi anemia, Schrader syndrome, Costerman syndrome, or any other known bone marrow failure syndrome;
4. A history of allogeneic stem cell transplantation;
5. Heart disease with grade III-IV heart failure [New York Heart Association (NYHA) classification] or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other clinically significant cardiac conditions within the year prior to enrollment;
6. The presence of any indwelling catheter or drainage tube (e.g., percutaneous nephrostomy tube, bile drainage tube or pleural/peritoneal/pericardial catheter), allowing the use of a dedicated central venous catheter;
7. Subjects with a history of CNS lymphoma, cerebrospinal fluid malignant cells or brain metastasis;
8. A history or disease of the central nervous system, such as seizure disorder, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving CNS;
9. The results of any of the following virology-ELISA tests were positive: HIV antibody, HCV antibody, TPPA, hepatitis B surface antigen;
10. There were active infections requiring systematic treatment within 2 weeks before single collection;
11. Persons with a known severe allergic reaction to cyclophosphamide or fludarabine, or with an allergic constitution;
12. A history of an autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that has caused injury to the terminal organs or requires systemic immunosuppressive/disease-modulating drugs within the past 2 years;
13. Pulmonary fibrosis is present;
14. Has received treatment in another clinical trial within 4 weeks prior to participation in this trial, or the date of signing of the informed consent is within 5 half-lives (whichever is longer) of the last medication used in the last other clinical trial;
15. Poor compliance due to physiological, family, social, geographical and other factors, unable to comply with the research program and follow-up plan;
16. The presence of a comorbiditie requiring systemic corticosteroid therapy (≥5 mg/ day of prednisone or equivalent dose of other corticosteroids) or other immunosuppressive agents within 6 months of study treatment was determined by the investigator;
17. Lactating women who do not want to stop breastfeeding;
18. Any other condition that the researcher considers inappropriate to be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within 28 days after cell infusion
  Proportion of patients with dose limiting toxicity (DLT) after cell infusion
Incidence of treatment-emergent adverse events (TEAEs) | 24 months after cell infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate(ORR) | Month 1,3,6,12,18and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 1,3,6,12,18and 24
Progression-free survival (PFS) | Month 6,12,18and 24
  Assessment of PFS at Month 6,12,18and 24
Overall survival (OS) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24
Duration of response(DOR) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No